CLINICAL TRIAL: NCT00001269
Title: Phase I Trial of FLAC (5-Fluorouracil, Leucovorin, Adriamycin, Cytoxan) Plus GM-CSF (Granulocyte-Macrophage Colony Stimulating Factor) Plus Dose Escalation of IL-3 (Interleukin-3) in Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910121; 91-C-0121
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Dose-Intensive Chemotherapy; Hematopoietic Growth Factor; Peripheral Blood Progenitor Cell
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Interleukin-3

INTERVENTIONS:
Drug: IL-3

SUMMARY:
This is a phase I study to determine the maximal tolerated dose of IL-3 given alone or sequentially with GM-CSF following FLAC chemotherapy in metastatic breast cancer patients.

DETAILED DESCRIPTION:
Phase I study to determine the maximal tolerated dose of IL-3 given alone or sequentially with GM-CSF following FLAC chemotherapy.

ELIGIBILITY:
Patients with Stage IV (metastatic) breast cancer are eligible who have a histologically-proven diagnosis. Measurable disease is not a prerequisite. Patients with Stage III disease or Stage ll with 7 or more nodes positive are eligible.

Patients who have had prior adjuvant chemotherapy and/or hormonal therapy are eligible providing the regimen did not include adriamycin. Patients who have had prior radiation therapy may be eligible providing there was not extensive radiation to the cardiac area or to greater than 20% of the bone marrow.

Patients who have received greater than 360mg/m2 of adriamycin as adjuvant therapy are ineligible.

Patient must be previously untreated with chemotherapy for metastatic disease.

There must be no history of previous malignancy except for cured non-melanoma skin cancer (basal or squamous cell carcinoma), cervical cancer in situ, or a past malignancy that has been inactive for over 5 years.

Performance status (Karnofsky scale) must be greater than 70; ECOG 0-2.

Absolute granulocyte count greater than 1500/mm3 and platelet count greater than 100,000/mm3.

Liver function tests (SCOT, Alk, Phosph., and T. Bili) should be less than 1.5 time the upper limits of normal. Serum creatinine should be less than 1.7 or creatinine clearance should be greater than 45 ml/min unless these abnormalities are due to tumor involvement.

The patient must be able to give an informed consent, and to return to NCI for treatment and adequate follow-up for the period the protocol requires.

No pregnant patients may be entered on this study; all patients should be informed about the need for contraception.

Patients must be greater than or equal to 18 years of age.

No patients who are poor medical or psychiatric risks because of nonmalignant systemic disease which would preclude them from being subjected to any treatments in this protocol.

No patients with a history of cardiac disease must have a normal ejection fraction by MUGA Scan and have no angina. Patients who have received prior adriamycin must have a LVEF greater than 45%.

No history of CNS metastasis, or known seizure disorder.

No allergy to any study medication.

No pregnant or lactacting women.

No patients requiring ongoing therapy for asthma.

No patients with bleeding disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1991-05; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Antman K, Gale RP. Advanced breast cancer: high-dose chemotherapy and bone marrow autotransplants. Ann Intern Med. 1988 Apr;108(4):570-4. doi: 10.7326/0003-4819-108-4-570. PMID 3279894
- [Background] Clark SC, Kamen R. The human hematopoietic colony-stimulating factors. Science. 1987 Jun 5;236(4806):1229-37. doi: 10.1126/science.3296190.
- [Background] Metcalf D, Begley CG, Johnson GR, Nicola NA, Vadas MA, Lopez AF, Williamson DJ, Wong GG, Clark SC, Wang EA. Biologic properties in vitro of a recombinant human granulocyte-macrophage colony-stimulating factor. Blood. 1986 Jan;67(1):37-45. PMID 3484428